CLINICAL TRIAL: NCT01673503
Title: A Prospective Study of Femtosecond Laser Intracorneal Lensectomi in Treatment of Moderate to High Myopia
Brief Title: A Prospective Study of Femtosecond Laser Intracorneal Lensectomi
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Anders H. Vestergaard, MD, PhD student, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20100111
Record Dates: First submitted 2012-08-20; First posted 2012-08-28 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Myopia; Astigmatism
Keywords: Myopia; refractive surgery; all femtosecond laser; ReLEx flex; ReLEx smile
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carl Zeiss Meditech VisuMax laser - ReLEx flex (Active Comparator): >30 patients will receive treatment for myopia with a VisuMax femtosecond laser from Carl Zeiss. The laser can cut with two different settings, called ReLEx flex and ReLEx smile. One eye will recieve ReLEx flex, and the other ReLEx smile
  Interventions: Device: Carl Zeiss Meditech VisuMax laser
- Carl Zeiss Meditech VisuMax laser - ReLEx smile (Active Comparator): >30 patients will receive treatment for myopia with a VisuMax femtosecond laser from Carl Zeiss. The laser can cut with two different settings, called ReLEx flex and ReLEx smile. One eye will recieve ReLEx flex, and the other ReLEx smile
  Interventions: Device: Carl Zeiss Meditech VisuMax laser

INTERVENTIONS:
Device: Carl Zeiss Meditech VisuMax laser — Refractive lenticule extraction (ReLEx) with the Carl Zeiss Meditech VisuMax laser
  Other Names: Refractive lenticule extraction, ReLEx

SUMMARY:
The purpose of this study is to compare visual acuity, safety, predictability, corneal biomechanics, dry eyes, and nerve-morphology after all femtosecond laser refractive lenticule extraction. Approximately 30 to 40 patients with moderate to high myopia will randomly (after ocular dominance) receive ReLEx flex in one eye, and ReLEx smile in the other.

ELIGIBILITY:
Inclusion Criteria:

* 25 to 45 years,
* moderate to high myopia with astigmatism =< 2 D,
* otherwise eye healthy,
* CDVA of 0.8 or better (Snellen).

Exclusion Criteria:

* systemic or ocular disease or previous eye surgery,
* thin cornea,
* a difference of more than 2 D myopia in the eyes of each subject.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35
Dates: Start 2011-05

PRIMARY OUTCOMES:
Visual acuity | up to 6 months
  Using ETDRS charts, both uncorrected and corrected distance visual acuity, along with visual acuity using the FrACT contrast chart

SECONDARY OUTCOMES:
refractive predictability | Pre-surgery, 1 week, 1 month, 3 months, 6 months
  Optometrists measure refraction at follow-up-examinations, and the refraction 6 monhts after surgery will be compared to the target refraction to calculate refractive predictability

OTHER OUTCOMES:
Corneal biomechanics, corneal nerve changes and dry eye symptoms | pre-surgery and 6 months after
  Corneal hysteresis and corneal resistence factor using the Ocular response analyser, nerve changes using the Cochet-Bonnet Aesthesiometer and confokal mikroscopy, and dry eyes symptoms using Schirmers test, Tear BUT, and Oculus keratograph, along with anterior segment OCT to measure tear meniscus hight.

CONTACTS AND LOCATIONS:
Overall Officials: Anders H Vestergaard, MD, Principal Investigator — Odense University Hospital, University of Southern Denmark
Locations (1):
- Department of Ophthalmology Aarhus Sygehus - Aarhus University Hospital, Denmark, Aarhus, Denmark

REFERENCES:
- [Derived] Vestergaard AH, Gronbech KT, Grauslund J, Ivarsen AR, Hjortdal JO. Subbasal nerve morphology, corneal sensation, and tear film evaluation after refractive femtosecond laser lenticule extraction. Graefes Arch Clin Exp Ophthalmol. 2013 Nov;251(11):2591-600. doi: 10.1007/s00417-013-2400-x. Epub 2013 Jun 22. PMID 23793872